CLINICAL TRIAL: NCT04192760
Title: Bifurcations Bad Krozingen (BBK) 3 - Trial Randomised Comparison of Culotte-stenting Versus DK-Crush--stenting for the Treatment of de Novo Non-left Main Coronary Bifurcation Lesions With Everolimus-eluting Stents
Brief Title: Culotte Versus DK-CRUSH Technique in Non-left Main Coronary Bifurcation Lesions
Acronym: BBK-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Principal Investigator, Dr. Miroslaw FERENC, Director of interventional cardiology department, University Heart Center Freiburg - Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHZ Bad Krozingen-cathlab
Record Dates: First submitted 2019-11-27; First posted 2019-12-10 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Coronary Stenosis; Stent Stenosis
Keywords: PCI; stent; bifurcation; Culotte; DK-Crush; restenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culotte Technique (Active Comparator): Both vessels have to be wired. Lesion preparation in the main vessel and side branch may be undertaken according to operator preference. After lesion preparation, the side branch has to be stented first. The first stent is placed from main branch into the side branch, covering the entire diseased segment with a wire jailed in the main vessel. The main vessel is rewired through the stent struts, and after removal of the jailed wire, is dilated with a balloon to separate stent struts. The side branch wire is then removed and the main vessel is stented covering the proximal and distal segment. The side-branch is re-wired and high pressure individual inflations are made in each vessel at the bifurcation point to ensure good stent strut separation. Afterwards, a lower pressure kissing inflation is made. Balloon sizing should be in accordance with the diameter of the vessel itself. Finally, a proximal optimization (POT) procedure is performed.
  Interventions: Procedure: Stenting
- DK-Crush Technique (Active Comparator): Both vessels have to be wired first. Lesion preparation in the main vessel and side branch may be undertaken according to operator preference (rotablation, if needed).
  After lesion preparation, the side branch is stented first. Side branch stent should have a small protrusion into the main branch. Before stent implantation in the side branch, an adequately sized balloon should be placed in the main branch, just opposite to the side branch ostium. After stent implantation in the side branch, stent balloon and wire are removed and the balloon in the main branch must be inflated, to crush the struts into the vessel wall. In next step, the new wire should be crossed into the ostium of the side branch and first kissing balloon dilatation will follow. The next step is to implant the second stent into the main branch, followed by second re-wiring, a second kissing balloon-dilatation and final proximal optimization (POT) procedure (single short balloon inflation in proximal segment).
  Interventions: Procedure: Stenting

INTERVENTIONS:
Procedure: Stenting — Comparison of two technical approaches in the interventional treatment on de-novo non-left main coronary lesions

SUMMARY:
Randomised comparison of Culotte technique versus "Double Kissing" - Crush technique (DK-Crush) for the percutaneous treatment of de novo non-left main coronary bifurcation lesions with modern everolimus-eluting stents (DES) - German multicenter study

DETAILED DESCRIPTION:
Aim of study This prospective randomized multicenter study will compare the long-term safety and efficacy of Culotte stenting versus "Double Kissing" - Crush (DK-Crush) stenting in the treatment of the de-novo non-left main coronary bifurcation lesions with new generation everolimus-eluting stents.

Study hypothesis In large coronary bifurcation lesions (main vessel > 2.5mm, side branch > 2.25mm) including significant ostial side branch disease, Culotte stenting compared with DKcrush stenting reduces maximal percent diameter stenosis at the bifurcation at 9-month follow-up by 25 %.

Study design Prospective, randomized, German multicenter study.

Methods Four-hundred patients, in whom a double-stenting technique is intended for the treatment of a non-left main de-novo coronary bifurcation lesion will be randomly assigned to Culotte stenting or to DK-crush stenting with an approved drug-eluting stent (SYNERGY-Stent). As a part of usual care, patients will undergo 9-month angiographic follow-up with quantitative coronary angiography. Clinical follow-up is planned at 1 year if no angiographic follow-up is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication, evidenced by angina / angina-equivalent symptoms or documented ischemia (non-invasive imaging such as scintigraphy, stress-MRI or stress-echo; FFR or iwFR) or patients with acute coronary syndromes (NSTE-ACS).
2. Clinical indication to perform double stenting only with Synergy™ stents for a clinically significant bifurcation stenosis as judged by the operator.
3. De-novo non-Ieft main coronary bifurcation lesions - 1,1,1 or 0,1,1 according to the Medina classification - of a native coronary artery with the following reference vessel diameters: main branch > 2,5 mm; side branch > 2,25 mm. The difference between vessel diameter of the main and side branch is ≤ 1 mm.
4. The target lesion has not been previously treated with any interventional procedure.
5. The target vessel (main branch and side branch) must appear feasible for stent implantation.
6. Patient has no other coronary intervention planned within 30 days of the procedure.
7. Patient has been informed of the nature of the study and agrees to its provisions and has written informed consent as approved by the Ethics Committee.
8. Patient is willing to comply with all required post-procedure follow-up.

Exclusion Criteria:

1. Patient had an acute ST-elevation myocardial infarction within 72 h preceding the index procedure or target vessel contains intraluminal thrombus.
2. Use of any other coronary stent than Synergy™ and Synergy Megatron™ except for baiI-out situations.
3. Patient with a known hypersensitivity or contraindication to the needed antithrombotic therapy, stent type or contrast media that cannot be adequately pre-medicated.
4. Non successful treatment of other lesion during the same procedure.
5. Patient with a severe bleeding diathesis, history of recent major bleeding or stroke (≤ 6 months), coagulopathy or severe liver disease.
6. Patient has a co-morbidity (i.e. cancer) that may cause the patient to be noncompliant with the protocol, or is associated with limited life-expectancy (Iess than 1 year).
7. Patient is participating in any other clinical study with an investigational product.
8. Patient is known to be pregnant or lactating at time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Angiographic restenosis in the bifurcation lesion by quantitative coronary analysis (QCA) | 9 months post index percutaneous coronary intervention (PCI)
  For quantitative coronary angiography, changes between result at the completion of the index intervention and at 9 months follow-up will be analysed using a computer based system dedicated to bifurcation analysis, according to the standard operating procedure of the angiographic core laboratory.
  Quantitative angiographic measurements will be obtained of the three segments of the bifurcation lesion: the proximal and distal segment of the main branch and the side branch. We will perform measurements in the stented portion of the vessel (in-stent) and in the distal or proximal 5 mm margin (edge). In-segment analyses will comprise the in-stent and the edge area.
  In addition, the bifurcation angle from the analysis system will be estimated.

SECONDARY OUTCOMES:
Incidence of target lesion revascularisation (TLR) | 1 year
  Any revascularisation (Re-PCI or CABG) at segments treated during index procedure
Incidence of major adverse cardiac events (MACE) | 1 year
  MACE defined as death, Myocardial infarction (Q wave and Non-Q wave), emergent cardiac bypass surgery, or TLR
Incidence of binary restenosis at any segment of the bifurcation lesion | 9 months
  ≥ 50% diameter stenosis in the main and side branch
Incidence of binary restenosis in the main and side branch | 9 months
  ≥ 50% diameter stenosis in main and side branch
Incidence of stent thrombosis (ST) | 1 year
  Post-procedure thrombotic stent occlusion according to the Academic Research Consortium-criteria

OTHER OUTCOMES:
Rate of device success | 9 months
  Attainment of < 30% residual stenosis of the target lesion in the main and side branch
Mean procedure time | Index Intervention
  Procedure time measured in minutes
Mean radiation exposure | Index Intervention
  Radiation exposure measured in cGym²
Mean volume of used contrast medium | Index Intervention
  Contrast medium measured in milliliters

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (13):
  - University Heart Center Freiburg • Bad Krozingen, Bad Krozingen, Suedring 15
  - Herz-u. Diabeteszentrum, Bad Oeynhausen
  - Herz-und Gefäßzentrum, Bad Segeberg
  - St. Johannes-Hospital, Dortmund
  - Herzzentrum Dresden an der Technischen Universität, Dresden
  - Elisabeth Krankenhaus, Essen
  - Universitätsklinikum Gießen, Giessen
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinik Mannheim, Mannheim
  - Deutsches Herzzentrum, München
  - Klinikum Oldenburg, Oldenburg
  - Herzzentrum Trier, Trier
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferenc M, Gick M, Comberg T, Rothe J, Valina C, Toma A, Loffelhardt N, Hochholzer W, Riede F, Kienzle RP, Achtari A, Neumann FJ. Culotte stenting vs. TAP stenting for treatment of de-novo coronary bifurcation lesions with the need for side-branch stenting: the Bifurcations Bad Krozingen (BBK) II angiographic trial. Eur Heart J. 2016 Dec 1;37(45):3399-3405. doi: 10.1093/eurheartj/ehw345. Epub 2016 Aug 30. PMID 27578807
- [Result] Chen SL, Xu B, Han YL, Sheiban I, Zhang JJ, Ye F, Kwan TW, Paiboon C, Zhou YJ, Lv SZ, Dangas GD, Xu YW, Wen SY, Hong L, Zhang RY, Wang HC, Jiang TM, Wang Y, Sansoto T, Chen F, Yuan ZY, Li WM, Leon MB. Clinical Outcome After DK Crush Versus Culotte Stenting of Distal Left Main Bifurcation Lesions: The 3-Year Follow-Up Results of the DKCRUSH-III Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1335-1342. doi: 10.1016/j.jcin.2015.05.017. PMID 26315736
- [Result] Chen SL, Zhang JJ, Ye F, Chen YD, Lu SZ, Tan H, Patel T, Kenji K, Tamari I, Shan SJ, Zhu ZS, Lin S, Tian NL, Li XB, Liu ZZ, Lee M, Wei M, Xu YW, Yuan ZB, Qian J, Sun XW, Yang S, Chen JG, He B, Sumit S. [Comparison of DK crush with classical crush technique with drug-eluting stents for the treatment of coronary bifurcation lesions from DKCRUSH-1 study]. Zhonghua Xin Xue Guan Bing Za Zhi. 2008 Feb;36(2):100-7. Chinese. PMID 19099943
- [Result] Chen SL, Santoso T, Zhang JJ, Ye F, Xu YW, Fu Q, Kan J, Paiboon C, Zhou Y, Ding SQ, Kwan TW. A randomized clinical study comparing double kissing crush with provisional stenting for treatment of coronary bifurcation lesions: results from the DKCRUSH-II (Double Kissing Crush versus Provisional Stenting Technique for Treatment of Coronary Bifurcation Lesions) trial. J Am Coll Cardiol. 2011 Feb 22;57(8):914-20. doi: 10.1016/j.jacc.2010.10.023. PMID 21329837
- [Result] Erglis A, Kumsars I, Niemela M, Kervinen K, Maeng M, Lassen JF, Gunnes P, Stavnes S, Jensen JS, Galloe A, Narbute I, Sondore D, Makikallio T, Ylitalo K, Christiansen EH, Ravkilde J, Steigen TK, Mannsverk J, Thayssen P, Hansen KN, Syvanne M, Helqvist S, Kjell N, Wiseth R, Aaroe J, Puhakka M, Thuesen L; Nordic PCI Study Group. Randomized comparison of coronary bifurcation stenting with the crush versus the culotte technique using sirolimus eluting stents: the Nordic stent technique study. Circ Cardiovasc Interv. 2009 Feb;2(1):27-34. doi: 10.1161/CIRCINTERVENTIONS.108.804658. Epub 2009 Feb 10. PMID 20031690
- [Result] Ferenc M, Buettner HJ, Gick M, Comberg T, Rothe J, Khoury F, Valina C, Toma A, Kuebler P, Riede F, Neumann FJ. Clinical outcome after percutaneous treatment of de novo coronary bifurcation lesions using first or second generation of drug-eluting stents. Clin Res Cardiol. 2016 Mar;105(3):230-8. doi: 10.1007/s00392-015-0911-7. Epub 2015 Sep 2. PMID 26329585
- [Result] Lee JM, Hahn JY, Kang J, Park KW, Chun WJ, Rha SW, Yu CW, Jeong JO, Jeong MH, Yoon JH, Jang Y, Tahk SJ, Gwon HC, Koo BK, Kim HS. Differential Prognostic Effect Between First- and Second-Generation Drug-Eluting Stents in Coronary Bifurcation Lesions: Patient-Level Analysis of the Korean Bifurcation Pooled Cohorts. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1318-1331. doi: 10.1016/j.jcin.2015.05.014. PMID 26315734

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04192760/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04192760/SAP_001.pdf